CLINICAL TRIAL: NCT04302584
Title: Comparison of Between Norepinephrine Alone Versus Norepinephrine / Vasopressin Combination for Resuscitation in Septic Shock
Brief Title: Norepinephrine / Vasopressin Combination for Resuscitation in Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hanaa Mohamed Abdallah ElGendy MD, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMASU MD 239/2016
Record Dates: First submitted 2020-02-28; First posted 2020-03-10 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Septic Shock; Acute Kidney Injury
MeSH Terms: conditions — Shock, Septic; Acute Kidney Injury | interventions — Norepinephrine; Vasopressins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NE (Active Comparator): patients received IV Norepinephrine infusion starting with (0.1mcg/kg/min)
  Interventions: Drug: norepinephrine / Vasopressin
- NE/VP (Active Comparator): patients received IV Norepinephrine infusion (Starting with (0.1 mcg/kg/min). +Vasopressin infusion at the rate of (0.03 unit/min)
  Interventions: Drug: norepinephrine / Vasopressin

INTERVENTIONS:
Drug: norepinephrine / Vasopressin — • The drug infusion was prepared as 100 IU of AVP (Pressyn; Ferring Inc., Toronto, Ontario, Canada) in 250 ml D5W, infused at the rate of 4.5 ml/h for 0.03 IU/min and 15 mg of Norepinephrine (Arterenol; Sanofi-Aventis, Frankfurt, Germany) in 250 ml D5W infused at the rate of 10 ml/h for 10 mcg/min using infusion pump.
  Other Names: norepinephrine

SUMMARY:
Although norepinephrine is commonly used and is the recommended agent for the treatment of hypotension in volume-resuscitated hyperdynamic septic shock, Low doses of vasopressin may be added to norepinephrine to maintain arterial blood pressure in refractory septic shock and to decrease exposure to norepinephrine. The aim of the work is to compare the effect of norepinephrine alone and Norepinephrine/vasopressin combination on hemodynamics and tissue perfusion in septic shock patients.

DETAILED DESCRIPTION:
Study which was performed on 90 adult of either sex in intensive care unit who developed septic shock.45 patients in each group according to the drugs used, by the single blind technique as the treating physician only is aware of the drugs used.

Group 1: patients received IV Norepinephrine infusion starting with (0.1mcg/kg/min).

Group 2: patients received IV Norepinephrine infusion (Starting with (0.1 mcg/kg/min). +Vasopressin infusion at the rate of (0.03 unit/min).

A comparison was done between both groups as regard:Hemodynamics,Tissue perfusion, C-Reactive Protein (mg/L) ,WBC, UREA (mg/dL),CREATININE (mg/dl), NGAL (Neutrophil gelatinase associated Lipocalin) (ng/ml). Comparison was done at baseline, then every 6 hours for 48 h as regard hemodynamics and tissue perfusion, and at base line then, 24 h and 48 h as regard sepsis biomarkers and renal biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years of both sex

Exclusion Criteria

* Patients with renal impairment (Creatinine>2mg/dl)
* Sever Heart Disease (ischemic/valvular)
* Peripheral vascular disease (e.g. Raynaud's phenomenon)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-05 (Actual); Study Completion 2019-01-06 (Actual)

PRIMARY OUTCOMES:
Lactate Level Lactate level • (central venous oxygen saturation)SVO2 | 48 hours
  mmol/L
Scvo2 | 48 hours

SECONDARY OUTCOMES:
NGAL, NGAL NGAL | 48 hours
  ng/ml
Mortality | 28 days
  28 days mortality
CRP | 48 hours
  mg/dl

CONTACTS AND LOCATIONS:
Locations (1):
- Hanaa El Gendy, Cairo, Ain Shams University Specialized Hospital, Egypt

IPD SHARING:
Plan to Share IPD: No